CLINICAL TRIAL: NCT01711138
Title: Active Streets, Active People - Junior: An Integrated Community Partnership to Enhance Physical Activity and Active Transport to School in Children and Youth
Brief Title: An Intervention Study to Assess the Role of the Built Environment on Physical Activity and Active Transportation to School in Children and Youth
Acronym: ASAP-Jr
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: City of Vancouver (Unknown); Vancouver School Board (Unknown); JW Sporta (Unknown); City of Surrey (Unknown); Surrey School Board (Unknown)
Responsible Party: Principal Investigator, Heather McKay, Principal Investigator, University of British Columbia
Other Study IDs: H12-01439
Record Dates: First submitted 2012-10-15; First posted 2012-10-22 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Physical Activity
Keywords: Physical Activity; Physical Fitness; Transportation; Environment Design; Child; Adolescent
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention: Intervention group is geographically located near a built environment intervention (neighbourhood redevelopment).
- Comparison: Comparison group is not exposed to the built environment intervention according to their geographic location.

SUMMARY:
The purpose of this study is to evaluate if changes to the built environment influence physical activity and active transport to school in children and youth.

ELIGIBILITY:
Inclusion Criteria:

* Student is in grade 4 - 10 at start of study (fall 2012), or grade 4 at any of the subsequent study years (2013-2015).
* Student's parent(s) or guardian(s) provide(s) consent.

Exclusion Criteria:

* Student is not in grade 4 - 10 at start of study (fall 2012).
* Student's parent(s) or guardian(s) do(es) not provide consent.
* Student cannot read or write in English.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants who attend school grades 4-10 at baseline (Fall 2012) will be invited to participate (intervention group). Participants (n-matched) who attend school grades 4-10 at baseline (Fall 2012) in a neighbouring catchment boundary will be invited to participate (comparison group).
Sampling Method: Non-Probability Sample
Enrollment: 573 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Objectively measured physical activity overall (minutes of moderate-to-vigorous physical activity per day) | up to 3 years
  Accelerometry (ActiGraph, FL, USA)

SECONDARY OUTCOMES:
Objectively measured physical activity during commuting to and from school (minutes of moderate-to-vigorous physical activity during commuting) | up to 3 years
  Accelerometry (ActiGraph, FL, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A McKay, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver, British Columbia, Canada